CLINICAL TRIAL: NCT04989101
Title: Nigelle 5 Study Project/ Prevention of Influenza Syndroms
Brief Title: Nigelle 5 in Prevention of Influanza
Acronym: NigCOV3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, PROFESSOR, Hôpital Universitaire Sahloul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NigCOV 3
Record Dates: First submitted 2021-07-24; First posted 2021-08-04 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: Nigelle 5CH; Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nigelle Group (Active Comparator): The candidate must take one capsule / day of nigella 5 for 21 days (1 bottle). Follow-up should be done weekly for 1 month.
  Interventions: Drug: Nigella
- Placebo Group (No Intervention): Follow-up should be done weekly for 1 month.

INTERVENTIONS:
Drug: Nigella — The candidate must take one capsule / day of nigella 5 for 21 days (1 bottle). Follow-up should be done weekly for 1 month.
  Arms: Nigelle Group

SUMMARY:
This study will be carried out by more than 30 liberal Tunisian doctors, who will submit according to the inclusion / exclusion criteria of people who will receive (free of charge) a capsule of the Nig5 product sublingually, each day. Against a control group which will be followed with the same protocol as the first but which will not receive the product. Randomization (even days: nigella group, odd days: control group)

DETAILED DESCRIPTION:
This study will focus on the evaluation of the natural product Nigella Sativa in the fractalized form. "Lactose Nigelle 5" from the Tunisian company Fractal Tun, in terms of possible contribution to the prevention of influenza-like illnesses, in particular COVID-19

It will be carried out by more than 30 liberal Tunisian doctors, who will submit according to the inclusion / exclusion criteria of people who will receive (free of charge) a capsule of the Nig5 product sublingually, each day. Against a control group which will be followed with the same protocol as the first but which will not receive the product. Randomization (even days: nigella group, odd days: control group)

The monitoring and evaluation will last for 3 weeks with taking the product Nig5, followed by a week without taking the product. That is 4 weeks in all.

More than 30 physicians volunteered to participate in this study without remuneration and without consultation fees for the candidates.

This study will be supervised by Professor Riadh Boukef, head of emergency services at Sahloul University Hospital, who will collect all the data afterwards in order to submit them to the statistical tools in force.

Professor Boukef will be responsible for preparing the abstract and publishing it on his behalf in the scientific journals of his choice, naming the doctors who participated as well as the product in question and the company that markets it in Tunisia.

27 free practice doctors participate in patient recruitment: AMICHE Sondèss BAHA Mohamed BEN AMARA Mohamed Khalil BEN ARBIA Karima BEN AYAD Afef BEN AYED KTARI Fouzia BENTALEB Mourad BESBES Mohamed CHTOUROU Iteb DHOUIB Manel DJAIT Mohamed DJEMAL Najla ELFIDHA Mongi FOURATI Imen FRIH Sabria FRIKHA Fahmi GHARBI Nadia KAMMOUN Naziha KETATA Mourad MHIRI Ikram NJAH Jamil OUARGHI Sameh REGAIEG Mourad SAKKA Samar TRABELSI Hinda ZOUARI Imen ZOUARI Nassira

ELIGIBILITY:
Inclusion Criteria:

* patients with an age> 40 years

Exclusion Criteria:

* Being positive for COVID or having contracted it previously
* Positive for COVID between D1 and D5 of the study, meaning that there was infection before inclusion.
* Immunocompromised (HIV, other ...)
* Under chemotherapy
* On immunosuppressants
* Pregnant women

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
SarsCOV2 Infection | one month
  Respiratory infection

SECONDARY OUTCOMES:
Contamination | one month
  contamination of the entourage in the event of respiratory infection by COVID19

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Sousse, Tunisia
Locations (1):
- HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Data Statistical analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available after publication
Access Criteria: all Criteria will be shared in the accepted article